CLINICAL TRIAL: NCT01665573
Title: Cannabinoid Augmentation of Fear Response in Humans
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Mohini Ranganathan, Assistant Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 120303009906
Record Dates: First submitted 2012-07-11; First posted 2012-08-15 (Estimated); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Fear Conditioning
Keywords: Fear Conditioning; Cannabinoids; Fear Response
MeSH Terms: interventions — N-pyridazin-3-yl-4-(3-((5-(trifluoromethyl)pyridin-2-yl)oxy)benzylidene)piperidine-1-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-04457845 (Active Comparator): Acquisition of conditioning Administration of drug Extinction of conditioning
  Interventions: Drug: PF-04457845; Drug: Placebo
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: PF-04457845; Drug: Placebo

INTERVENTIONS:
Drug: PF-04457845 — Acquisition of conditioning Administration of drug Extinction of conditioning
Drug: Placebo — Acquisition of conditioning Administration of placebo Extinction of conditioning

SUMMARY:
The purpose of this double blind, randomized, controlled, proof-of-concept study is to test the effects of cannabinoid receptor augmentation on the facilitation of fear conditioning. On three days over not more than two weeks, subjects will be trained to associate cues with two different stimuli, then this association will be extinguished. Cannabinoid receptor stimulation will be accomplished indirectly by harnessing the brain's capacity to endocannabinoids through the administration of an enzyme (FAAH inhibitor) that prevents degradation of anandamide. Subjects will receive placebo or the FAAH-inhibitor PF-04457845. Some details of this study have not been disclosed to preserve the study design.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 65
* Male and female
* No major medical problems

Exclusion Criteria:

* Hearing problems
* Psychiatric or mental problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-07-17 (Actual); Primary Completion 2015-10-16 (Actual); Study Completion 2015-10-16 (Actual)

PRIMARY OUTCOMES:
Galvanic skin response | Test days #1, #2, and #3, on average a week
  Measure of sympathetic autonomic activation
Cortisol levels measured in blood | Test days #1, #2, and #3, on average a week
  Salivary b-amylase and serum cortisol levels will be assessed as neurochemical measures of stress response.

CONTACTS AND LOCATIONS:
Overall Officials: Mohini Ranganathan, MD, Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States